CLINICAL TRIAL: NCT01895127
Title: Efficacy and Safety of Eculizumab for Treatment of Antibody-mediated Rejection Following Renal Transplantation.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Anil K. Chandraker, MD, Medical Director of Kidney and Pancreas Transplantation, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013P001292
Record Dates: First submitted 2013-06-28; First posted 2013-07-10 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-08

CONDITIONS: Antibody-mediated Rejection; Humoral Rejection
Keywords: Kidney Transplant; Renal Transplant; Rejection; Antibody mediated; Humoral; Eculizumab
MeSH Terms: conditions — Rejection, Psychology | interventions — eculizumab; Immunoglobulins; Immunoglobulins, Intravenous; Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (Active Comparator): * Plasmapheresis (PP) x 3, at 40-60 cc/kg.
  * Immunoglobulin (IVIg), to be administered after each PP
  Interventions: Biological: Immunoglobulin; Procedure: Plasmapheresis
- Soliris (eculizumab) (Experimental): * 1200 mg first dose (Time: Screening/Week "0", after Biopsy Proven AMR)
  * 900 mg weekly for 4 doses (Weeks 1, 2, 3, 4)
  * 1200 mg week 5
  * Week 6: If donor specific antibody < 50% of baseline DSA then no further treatment, otherwise 1200 mg weeks 7, 9
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab
  Other Names: Soliris
  Arms: Soliris (eculizumab)
Biological: Immunoglobulin
  Other Names: IVIg
  Arms: Standard of Care
Procedure: Plasmapheresis
  Arms: Standard of Care

SUMMARY:
This is an open-label analysis that will compare eculizumab versus Plasmapheresis (PP) and Immunoglobulin (IVIg) for the treatment of antibody-mediated rejection (AMR) in renal transplant recipients. All patients will be evaluated from the time of AMR diagnosis for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adult renal transplant recipients, men and women between 18 and 75 years of age.
2. Any patient with acute graft dysfunction (elevation of creatinine above post transplant nadir)

   AND, two out of three, of the following Inclusion Criteria:
3. Presence of circulating anti human leukocyte antigen (HLA) antibody (DSA "donor specific antibody").
4. Histological findings compatible with Banff Class II or III AMR on transplant biopsy.
5. Peritubular capillary c4d positivity on transplant biopsy.

Exclusion Criteria:

1. Patients that have received eculizumab prior to enrolling in the study.
2. Patients with ongoing non-acute antibody mediated rejection.
3. Patients with predominantly chronic antibody mediated rejection or interstitial fibrosis/tubular atrophy.
4. History of severe cardiac disease (e.g., New York Heart Association [NYHA] Functional Class III or IV, myocardial infarction ≤ 6 months of randomization, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina or other significant cardiovascular diseases)
5. Prior splenectomy
6. Has a known bleeding disorder
7. Has any active bacterial or other infection which is clinically significant in the opinion of the Investigator and is a contraindication to transplantation
8. Has participated in any other investigational drug study or was exposed to an investigational drug or device within 30 days of screening
9. Has received rituximab (Rituxan®) ≤ 3 months prior to screening
10. Has received bortezomib (Velcade®) ≤ 3 months prior to screening
11. Has received alemtuzumab (Campath®) ≤ 6 months prior to screening
12. Need for concurrent treatment with anti thymocyte globulin (Thymoglobulin®)
13. Hypersensitivity to murine proteins or to one of the product excipients
14. History of illicit drug use or alcohol abuse within the previous year
15. Unresolved meningococcal disease
16. Pregnancy or lactation
17. Current cancer or a history of cancer within the 5 years prior to screening with the exception of patients who have successfully treated non-metastatic basal or squamous cell carcinoma of the skin; carcinoma in situ of the cervix; or breast carcinoma in situ
18. Any medical condition that, in the opinion of the Investigator, might interfere with the patient's participation in the study, poses an added risk for the patient, or confounds the assessment of the patient Active infection with Hepatitis B (HBV), Hepatitis C (HCV) or human immunodeficiency virus (HIV)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anil K Chandraker, MD, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - UCSF Medical Center, San Francisco, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: * Plasmapheresis (PP) x 3, at 40-60 cc/kg.
  * Immunoglobulin (IVIg), to be administered after each PP
  Immunoglobulin
  Plasmapheresis
- Soliris (Eculizumab): * 1200 mg first dose (Time: Screening/Week "0", after Biopsy Proven AMR)
  * 900 mg weekly for 4 doses (Weeks 1, 2, 3, 4)
  * 1200 mg week 5
  * Week 6: If donor specific antibody < 50% of baseline DSA then no further treatment, otherwise 1200 mg weeks 7, 9
  Eculizumab
Period: Screening
Arm/Group | Standard of Care | Soliris (Eculizumab)
Started | 4 | 7
Completed | 4 (One subject was found to be pregnant at screening so was withdrawn from the study prior to treatment) | 7
Not Completed | 0 | 0
Period: Treatment Period (Week 0-Month 3)
Arm/Group | Standard of Care | Soliris (Eculizumab)
Started | 3 | 7
Completed | 3 | 7
Not Completed | 0 | 0
Period: Month 3 Follow-up & Biopsy
Arm/Group | Standard of Care | Soliris (Eculizumab)
Started | 3 | 7
Completed | 3 | 7
Not Completed | 0 | 0
Period: Long Term Follow-up (Month 3-12)
Arm/Group | Standard of Care | Soliris (Eculizumab)
Started | 3 | 7
Completed | 1 | 4
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Soliris (Eculizumab) | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 43.25 [24 to 61] | 43.29 [30 to 59] | 43.27 [24 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Estimated Glomerular Filtration (eGFR) Rate
Description: Percent change in eGFR rate at 3 months post-treatment using the modified Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
Time Frame: Month 3
Population: 1 subject in the SOC arm received rescue therapy, per protocol, with eculizumab following PP/IVIg. 1 subject in the Soliris arm received SOC therapy (PP/IVIg) following completion of Soliris treatment period. Both of these subjects received both SOC and Soliris treatment prior to Month 3 protocol biopsy so we have listed their outcome separately.
Measure: Mean (Full Range); unit: percent change in eGFR from wk 0 to mo 3
Groups:
- Standard of Care + Soliris (Eculizumab): Subjects received both standard of care and Soliris treatment between Week 0 and Month 3
Arm/Group | Standard of Care | Soliris (Eculizumab) | Standard of Care + Soliris (Eculizumab)
Number analyzed (Participants) | 2 | 6 | 2
percent change in eGFR from wk 0 to mo 3 | -12.92 [-13.33 to -12.5] | 12.60 [-34.29 to 136.36] | 377.25 [25.93 to 728.57]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the duration of the trial starting at screening through Month 12 for each subject.
Arm/Group | Standard of Care | Soliris (Eculizumab)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7
Serious Adverse Events (participants affected / at risk) | 3/4 | 5/7
Other Adverse Events (participants affected / at risk) | 3/4 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=4) | Soliris (Eculizumab) (N=7)
elevated serum alkaline phosphatase (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (2) — elevated creatinine, no biopsy to for additional diagnosis
Cellular Rejection (Immune system disorders) | 1 (1) | 3 (3) — biopsy proven
Antibody-mediated rejection (Immune system disorders) | 3 (4) | 5 (5) — biopsy proven, ongoing rejection
Hypertension (Cardiac disorders) | 0 | 1
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (3) | 0 (0)
Pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Bilateral Ear Infection (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=4) | Soliris (Eculizumab) (N=7)
headache (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Edema (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Emesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Fever (Infections and infestations) | 3 (5) | 2 (4)
Dizziness (General disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (2) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (2) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 0 (0) — increased creatinine
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1)
Cough (General disorders) | 1 (2) | 1 (1)
Hyperkalemia (General disorders) | 1 (1) | 0 (0)
elevated alkaline phosphatase (General disorders) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Back Pain (General disorders) | 1 (1) | 1 (1)
Insomnia (General disorders) | 1 (1) | 0 (0)
Weight Gain (General disorders) | 1 (1) | 1 (1)
Tremor (General disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No